CLINICAL TRIAL: NCT04515901
Title: Early Intervention Sphenopalatine Ganglion Blocks (SPGBs) Versus Standard Conservative Management of Post Dural Puncture Headache in Obstetric Patients - A Randomized Feasibility Study
Brief Title: Spenopalatine Ganglion Block for Treatment of Post-dural Puncture Headaches
Acronym: SPGB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll participants.
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7978
Record Dates: First submitted 2020-08-11; First posted 2020-08-17 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Postdural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPGB (Experimental): Via a soft tip 20-gauge long IV catheter attached to a 3 mL syringe will be filled with 2 mL of 2% viscous lidocaine. The 2% viscous lidocaine will be administered according to the method of Barre.
  Interventions: Drug: 2% lidocaine
- Placebo (Placebo Comparator): It will be adminstered the same as the experimental arm but with methylcellulose and cherry flavouring to match odour and taste.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 2% lidocaine — Viscous lidocaine
  Arms: SPGB
Other: Placebo — Methylcellulose and cherry flavouring
  Arms: Placebo

SUMMARY:
Postdural puncture headache (PDPH) is a severe, debilitating complication of dural puncture that can arise from insertion of an epidural or spinal needle for labour analgesia. Presently, the conservative treatment options for PDPH have limited effectiveness and the gold standard treatment for PDPH, an epidural blood patch, is an invasive intervention with the potential for serious complications. There is a growing number of case reports and retrospective studies that suggest a sphenopalatine ganglion block (SPGB) with local anesthetic may offer an effective, safe, and easy-to-administer treatment option for PDPH in postpartum patients. We aim to conduct a feasibility study to assess whether a randomized controlled trial is feasible comparing whether early intervention SPGB with the option for repeat, patient self-administered SPGBs versus current standard conservative management can reduce the severity and duration of PDPH pain and improve patient functional status.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* Confirmed PDPH as per ICHD-3 diagnostic criteria

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) class 4 and above
* History of chronic headaches or migraines requiring prescription medication
* Known nasal septal deformity or abnormality
* Known allergy to amide anesthetics
* Intrathecal catheters
* Patients who received EBP on the initial presentation with PDPH who declined a trial of conservative management
* Postpartum complication delaying maternal discharge

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Enrollment rate | 6 months
  Number of consented patients over number of number of eligible patients

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angle P, Tang SL, Thompson D, Szalai JP. Expectant management of postdural puncture headache increases hospital length of stay and emergency room visits. Can J Anaesth. 2005 Apr;52(4):397-402. doi: 10.1007/BF03016283. PMID 15814755
- [Background] Barre F. Cocaine as an abortive agent in cluster headache. Headache. 1982 Mar;22(2):69-73. doi: 10.1111/j.1526-4610.1982.hed2202069.x. No abstract available. PMID 7085264
- [Background] Channabasappa SM, Manjunath S, Bommalingappa B, Ramachandra S, Banuprakash S. Transnasal sphenopalatine ganglion block for the treatment of postdural puncture headache following spinal anesthesia. Saudi J Anaesth. 2017 Jul-Sep;11(3):362-363. doi: 10.4103/sja.SJA_59_17. No abstract available. PMID 28757848
- [Background] Choi PT, Galinski SE, Takeuchi L, Lucas S, Tamayo C, Jadad AR. PDPH is a common complication of neuraxial blockade in parturients: a meta-analysis of obstetrical studies. Can J Anaesth. 2003 May;50(5):460-9. doi: 10.1007/BF03021057. PMID 12734154